CLINICAL TRIAL: NCT03504774
Title: T Cell Reagent Research for Monitoring T Cells in Food Allergy (MOTIF) Phase 2 Study Using Food Allergen Oral Immunotherapy for Shrimp or Cashew Allergies
Brief Title: Food Allergen OIT for Shrimp and Cashew
Acronym: MOTIF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study discontinued due to slow enrollment during COVID-19 pandemic
Sponsor: Sayantani B. Sindher (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Sayantani B. Sindher, Sponsor Investigator, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-48330; 1U01AI140498-01 (NIH)
Record Dates: First submitted 2018-04-03; First posted 2018-04-20 (Actual); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Allergy;Food; Allergy to Shrimp; Allergy to Cashew Nut (Disorder)
Keywords: OIT; Oral Immunotherapy; Cashew Allergy; Shrimp Allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Food allergy OIT in a single group design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cashew or Shrimp Oral Immunotherapy (Experimental): Participants, ages 7 to 55 years, inclusive, with an allergy to Cashew or Shrimp.
  Interventions: Drug: Cashew or Shrimp Oral Immunotherapy

INTERVENTIONS:
Drug: Cashew or Shrimp Oral Immunotherapy — All cohorts will undergo an updosing regimen starting at 5 mg allergen, with dose escalation every 2 weeks to reach a 1000 mg dose at week 28, after which they will be maintained at that dose for 24 weeks. At the conclusion of the maintenance phase (Week 52), participants will undergo DBPCFC.
  Other Names: OIT

SUMMARY:
A prospective Phase 2, single-center, single-allergen OIT of cashew or shrimp in participants with proven allergies to either cashew or shrimp, respectively. We intend to treat 72 participants, ages 7 to 55 years with an allergy to either cashew, or shrimp determined by Double Blind-Placebo Controlled-Food Challenge (DBPCFC), allergy history, clinical symptoms, food-allergen (FA)-specific IgE levels, and skin prick test (SPT).

DETAILED DESCRIPTION:
A prospective Phase 2, single-center, single-allergen OIT of cashew or shrimp in participants with proven allergies to either cashew or shrimp, respectively. We intend to treat 72 participants, ages 7 to 55 years with an allergy to either cashew or shrimp determined by Double Blind-Placebo Controlled-Food Challenge (DBPCFC), allergy history, clinical symptoms, food-allergen (FA)-specific IgE levels, and skin prick test (SPT). Enrolled participants must be positive at or before the 300 mg (443 mg cumulative) dosing level of FA protein. OIT treatment groups will be cashew or shrimp.

All cohorts will undergo an updosing regimen starting at 5 mg allergen, with dose escalation every 2 weeks to reach a 1000 mg dose at week 28, after which they will be maintained at that dose for 24 weeks. At the conclusion of the maintenance phase (Week 52), participants will undergo DBPCFC. Participants that pass their food challenge with no or mild objective reactions to up to a cumulative 2043 mg of the FA allergen in their OIT at the end of this phase (primary outcome) will be considered desensitized and have successfully met the primary endpoint.

All participants then will continue in the study by undergoing withdrawal from OIT for 6 weeks to examine mechanisms underlying sustained responsiveness (SU) which will be defined as a participant's passing a DBPCFC with no or mild objective reaction to up to a cumulative 2043 mg of the FA allergen in their DBPCFC at week 58.

Those participants who pass the Week 58 challenge up to a cumulative of 2043 mg will be given the option to continue the withdrawal phase up to Week 64 which will be end of study. Week 58 will be end of study for those who do not opt for this continuation of withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or parent guardian must be able to understand and provide informed consent
* Age 7 through 55 years (inclusive)
* Clinical history of allergy to cashew or shrimp-containing foods
* Serum IgE to cashew or shrimp of ≥0.35 kUA/L [determined by UniCAPTM within the past 12 months] and/or a SPT to cashew or shrimp ≥3 mm compared to control
* Experience dose-limiting symptoms at or before the 300 mg challenge dose of FA protein on Screening DBPCFC conducted in accordance with PRACTALL guidelines
* Written informed consent from adult participants
* Written informed consent from parent/guardian for minor participants
* Written assent from minor participants as appropriate (e.g., above the age of 7 years or the applicable age per local regulatory requirements)
* All female subjects of child-bearing potential will be required to provide a blood or urine sample for pregnancy testing that must be negative one week before being allowed to participate in the study.
* Use of effective birth control by female participants of child-bearing potential.

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol
* History of uncontrolled cardiovascular disease, including uncontrolled hypertension
* History of other chronic disease (other than asthma, atopic dermatitis, or allergic rhinitis) requiring therapy (e.g., heart disease, diabetes) that is, or is at significant risk of becoming unstable or requiring a change in chronic therapeutic regimen and, in the opinion of the Principal Investigator, would represent a risk to the subject's health or safety in this study or the subject's ability to comply with the study protocol.
* History of eosinophilic esophagitis (EoE), other eosinophilic gastrointestinal disease, chronic, recurrent, or severe gastroesophageal reflux disease (GERD) grade 3 according to CTCAE version 5.0, symptoms of dysphagia (e.g., difficulty swallowing, food "getting stuck"), or recurrent gastrointestinal symptoms of undiagnosed etiology
* Current participation in any other interventional study
* Subject is currently in the build-up phase of immunotherapy to another allergen and is on maintenance immunotherapy dose for any allergen related to cashew or shrimp
* Severe asthma (NAEPP EPR-3 Medication Criteria Steps 5 or 6)
* Mild or moderate asthma (NAEPP EPR-3 Medication Criteria Steps 1-4), if not controlled as indicated by an ACT<19
* A hospitalization for asthma in the past 6 months
* ER visit for asthma within the past 6 months
* Burst or steroid course for asthma in the past 6 months
* Use of omalizumab or biologic therapy (e.g., infliximab, rituximab, etc.) within the past 6 months
* Use of complementary and alternative medicine (CAM) treatment modalities (e.g., herbal remedies) for atopic and /or non-atopic disease within 90 days preceding Initial Dose Escalation Day (IDED) or at any time after the IDED
* Use of beta-blockers (oral)
* Pregnancy or lactation
* Allergy to oat
* History of severe anaphylaxis to cashew or shrimp with symptoms including hypotension requiring fluid resuscitation and/or the need for mechanical ventilation within the last year
* Use of investigational drugs within 12 weeks of participation
* Past or current medical problems or findings from physical assessment or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study

Ages: 7 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sayantani Sindher, MD, Study Director — Stanford University, SNP Center for Food Allergy and Asthma Research
Locations (1):
- Sean N Parker Center For Allergy and Asthma Research, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sindher SB, Fernandes A, Manohar M, Cao S, Gupta S, Parsons E, Bogetic D, Kumar D, Rogers J, Thompson J, Dunham D, Do E, Maysel-Auslender S, Liu TA, Martinez K, Anderson B, Kaushik A, Desai M, Maecker H, Perry S, Wheatley LM, Nadeau KC, Chinthrajah RS. Trends in allergen-reactive CRTH2+ T cells and TARC associated with successful outcomes in a phase 2 cashew oral immunotherapy study. Front Immunol. 2025 Oct 22;16:1655975. doi: 10.3389/fimmu.2025.1655975. eCollection 2025. PMID 41200192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with an allergy to Cashew or Shrimp were enrolled. The study was to examine the efficacy of oral immunotherapy regimen overtime, without comparisons between allergen groups.
Pre-assignment Details: 58 participants consented and assessed for eligibility. 2 participants withdrew consent and 4 participants screen failed, and were not allocated to treatment.
Groups:
- Cashew Oral Immunotherapy: Participants, ages 7 to 55 years, inclusive, with an allergy to Cashew, received updosing regimen starting at 5 mg allergen, with dose escalation every 2 weeks to reach a 1000 mg dose at week 28, after which they will be maintained at that dose for 24 weeks. At the conclusion of the maintenance phase (Week 52), participants will undergo Double Blind-Placebo Controlled-Food Challenge (DBPCFC). After week 52, participants will avoid the allergen (withdrawal phase) for 6 weeks and will come back for DBPCFC at week 58.
- Shrimp Oral Immunotherapy: Participants, ages 7 to 55 years, inclusive, with an allergy to Shrimp, received an updosing regimen starting at 5 mg allergen, with dose escalation every 2 weeks to reach a 1000 mg dose at week 28, after which they will be maintained at that dose for 24 weeks. At the conclusion of the maintenance phase (Week 52), participants will undergo DBPCFC. After week 52, participants will avoid the allergen (withdrawal phase) for 6 weeks and will come back for DBPCFC at week 58.
Period: Overall Study
Arm/Group | Cashew Oral Immunotherapy | Shrimp Oral Immunotherapy
Started | 40 | 12
Enrolled for the Intention-to-Treat Analysis | 40 | 12
Assigned to Build-up and Maintenance | 40 | 12
Had Week 52 Desensitization DBPCFC | 27 | 8
Had Week 58 Sustained Unresponsiveness DBPCFC | 26 | 8
Completed | 26 | 8
Not Completed | 14 | 4
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 11 | 3
Not completed — failed wk 52 DBPCFC | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cashew Oral Immunotherapy: Participants with an allergy to Cashew.
- Shrimp Oral Immunotherapy: Participants with an allergy to Shrimp.
- Total: Total of all reporting groups
Arm/Group | Cashew Oral Immunotherapy | Shrimp Oral Immunotherapy | Total
Number analyzed (Participants) | 40 | 12 | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14 [11 to 15.25] | 23.5 [17.25 to 37.75] | 14 [13 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 8 | 27
  Male | 21 | 4 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 35 | 11 | 46
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 18 | 4 | 22
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 0 | 0
  White | 11 | 7 | 18
  More than one race | 9 | 0 | 9
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 12 | 52
History of Asthma [Count of Participants; unit: Participants] | 19 | 7 | 26
History of Allergic Rhinitis [Count of Participants; unit: Participants] | 28 | 9 | 37
History of Atopic Dermatitis [Count of Participants; unit: Participants] | 24 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Expression of CD28 in the CD4+ Allergen Specific (CD154+)
Description: Expression of CD28 in the CD4+ allergen specific (CD154+) T-cells at baseline and 52 weeks, reported as the percentage of allergen specific (reactive) cells.
Time Frame: baseline and 52 week
Population: participants with baseline and week 52 CD28 expression data
Measure: Median (Full Range); unit: percentage of allergen reactive cells
Groups:
- All Participants: Participants with allergy to Cashew / Shrimp
Arm/Group | Cashew Oral Immunotherapy | Shrimp Oral Immunotherapy | All Participants
Number analyzed (Participants) | 25 | 8 | 33
percentage of allergen reactive cells
  baseline | 99 [88.7 to 100] | 98.9 [88.7 to 100] | 99 [88.7 to 100]
  week 52 | 100 [95.5 to 100] | 97.7 [93.8 to 100] | 99.5 [93.8 to 100]
Statistical Analysis 1: Comparison: All Participants; analysis of the change from baseline in CD28 expression; Test type: Other; p = 0.30, Mixed Models Analysis; Mean Difference (Net) = 0.6

2. Secondary Outcome: Expression of CD28+ Allergen Specific (CD154+) T-cells
Description: Expression of CD28+ allergen specific (CD154+) T-cells at baseline, week 52, and week 58, reported as the percentage of allergen specific (reactive) cells.
Time Frame: baseline, week 52 and week 58
Population: participants with baseline, week 52, or week 58 CD28 expression
Measure: Median (Full Range); unit: percentage of allergen reactive cells
Arm/Group | Cashew Oral Immunotherapy | Shrimp Oral Immunotherapy | All Participants
Number analyzed (Participants) | 25 | 8 | 33
percentage of allergen reactive cells
  baseline | 99 [88.7 to 100] | 98.9 [88.7 to 100] | 99 [88.7 to 100]
  week 52 | 100 [95.5 to 100] | 97.7 [93.8 to 100] | 99.5 [93.8 to 100]
  week 58: number analyzed (Participants) | 24 | 8 | 32
  week 58 | 100 [93.8 to 100] | 99.2 [93 to 100] | 100 [93 to 100]
Statistical Analysis 1: Comparison: Cashew Oral Immunotherapy; within-group analysis of change from baseline to week 52; Test type: Other; p = 0.82, Mixed Models Analysis; Mean Difference (Net) = 0.9
Statistical Analysis 2: Comparison: Cashew Oral Immunotherapy; within-group analysis on the change from baseline to week 58; Test type: Other; p = 0.053, Mixed Models Analysis; Mean Difference (Net) = 1.2
Statistical Analysis 3: Comparison: Cashew Oral Immunotherapy; within-group analysis of change from week 52 to week 58; Test type: Other; p = 0.062, Mixed Models Analysis; Mean Difference (Net) = 0.3
Statistical Analysis 4: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change from baseline to week 52; Test type: Other; p = 0.30, Mixed Models Analysis; Mean Difference (Net) = 0.2
Statistical Analysis 5: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change from baseline to week 58; Test type: Other; p = 0.54, Mixed Models Analysis; Mean Difference (Net) = 1.0
Statistical Analysis 6: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change from week 52 to week 58; Test type: Other; p = 0.82, Mixed Models Analysis; Mean Difference (Net) = 1.2

3. Secondary Outcome: Expression of the Mechanistic Markers Vis Luminex Assay
Description: Expression of the following measures in CD4+CD28+ allergen specific (CD154+) T-cells at baseline, week 52, and week 58. Data were collected for IFN-gamma, IL-4 and IL-10 via Luminex assay. Data collection was planned for receptor diversity in allergen specific T cell CDR3b as compared to non-specific T cells, and TGF beta, but these data were not collected. The median value (with full range) of mean fluorescence intensity across participants is reported for each time point.
Time Frame: baseline, week 52, and week 58
Population: participants who had baseline, week 52, or week 58 Luminex data
Measure: Median (Full Range); unit: mean fluorescence intensity
Arm/Group | Cashew Oral Immunotherapy | Shrimp Oral Immunotherapy | All Participants
Number analyzed (Participants) | 27 | 8 | 35
mean fluorescence intensity
  IFN-gamma at baseline | 53 [42 to 134] | 53.8 [46 to 78] | 53 [42 to 134]
  IFN-gamma at week 52 | 56 [33.5 to 128] | 61.2 [47 to 100] | 60 [33.5 to 128]
  IFN-gamma at week 58: number analyzed (Participants) | 26 | 8 | 34
  IFN-gamma at week 58 | 53 [33 to 248] | 58 [44 to 72] | 55 [33 to 248]
  IL-4 at baseline | 33 [18 to 55] | 30.2 [26.5 to 41] | 32 [18 to 55]
  IL-4 at week 52 | 32 [15 to 74] | 34 [22 to 46.5] | 33 [15 to 74]
  IL-4 at week 58: number analyzed (Participants) | 26 | 8 | 34
  IL-4 at week 58 | 33.5 [18 to 86] | 30 [21.5 to 38.5] | 32.5 [18 to 86]
  IL-10 at baseline | 36.5 [21 to 52] | 36.5 [26 to 42] | 36.5 [21 to 52]
  IL-10 at week 52 | 38.5 [26.5 to 75] | 38.5 [26 to 46.5] | 38.5 [26 to 75]
  IL-10 at week 58: number analyzed (Participants) | 26 | 8 | 34
  IL-10 at week 58 | 37 [29 to 61] | 36.2 [25 to 55] | 37 [25 to 61]
Statistical Analysis 1: Comparison: Cashew Oral Immunotherapy; within-group analysis of change in INFG from baseline to week 52; Test type: Other; p = 0.25, Mixed Models Analysis; Mean Difference (Net) = 4.8
Statistical Analysis 2: Comparison: Cashew Oral Immunotherapy; within-group analysis of change in INFG from baseline to week 58; Test type: Other; p = 0.24, Mixed Models Analysis; Mean Difference (Net) = 10.8
Statistical Analysis 3: Comparison: Cashew Oral Immunotherapy; within-group analysis of change in INFG from week 52 to week 58; Test type: Other; p = 0.61, Mixed Models Analysis; Mean Difference (Net) = 6
Statistical Analysis 4: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change in INFG from baseline to week 52; Test type: Other; p = 0.034, Mixed Models Analysis; Mean Difference (Net) = 8.5
Statistical Analysis 5: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change in INFG from baseline to week 58; Test type: Other; p = 0.45, Mixed Models Analysis; Mean Difference (Net) = 0.8
Statistical Analysis 6: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change in INFG from week 52 to week 58; Test type: Other; p = 0.12, Mixed Models Analysis; Mean Difference (Net) = 7.7
Statistical Analysis 7: Comparison: Cashew Oral Immunotherapy; within-group analysis of change in IL4 from baseline to week 52; Test type: Other; p = 0.83, Mixed Models Analysis; Mean Difference (Net) = 1
Statistical Analysis 8: Comparison: Cashew Oral Immunotherapy; within-group analysis of change in IL4 from baseline to week 58; Test type: Other; p = 0.67, Mixed Models Analysis; Mean Difference (Net) = 2
Statistical Analysis 9: Comparison: Cashew Oral Immunotherapy; within-group analysis of change in IL4 from week 52 to week 58; Test type: Other; p = 0.80, Mixed Models Analysis; Mean Difference (Net) = 1
Statistical Analysis 10: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change in IL4 from baseline to week 52; Test type: Other; p = 0.46, Mixed Models Analysis; Mean Difference (Net) = 1.7
Statistical Analysis 11: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change in IL4 from baseline to week 58; Test type: Other; p = 0.48, Mixed Models Analysis; Mean Difference (Net) = 3.2
Statistical Analysis 12: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change in IL4 from week 52 to week 58; Test type: Other; p = 0.25, Mixed Models Analysis; Mean Difference (Net) = 3.2
Statistical Analysis 13: Comparison: Cashew Oral Immunotherapy; within-group analysis of change in IL10 from baseline to week 52; Test type: Other; p = 0.14, Mixed Models Analysis; Mean Difference (Net) = 2.6
Statistical Analysis 14: Comparison: Cashew Oral Immunotherapy; within-group analysis of change in IL10 from baseline to week 58; Test type: Other; p = 0.73, Mixed Models Analysis; Mean Difference (Net) = 0.6
Statistical Analysis 15: Comparison: Cashew Oral Immunotherapy; within-group analysis of change in IL10 from week 52 to week 58; Test type: Other; p = 0.16, Mixed Models Analysis; Mean Difference (Net) = 2
Statistical Analysis 16: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change in IL10 from baseline to week 52; Test type: Other; p = 0.47, Mixed Models Analysis; Mean Difference (Net) = 1.8
Statistical Analysis 17: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change in IL10 from baseline to week 58; Test type: Other; p = 0.84, Mixed Models Analysis; Mean Difference (Net) = 1.1
Statistical Analysis 18: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change in IL10 from week 52 to week 58; Test type: Other; p = 0.55, Mixed Models Analysis; Mean Difference (Net) = 0.7

4. Secondary Outcome: Expression of the Mechanistic Marker Via Flow Cytometry
Description: Expression of the following measures in CD4+CD28+ allergen specific (CD154+) T-cells at baseline, week 52, and week 58. Data were collected for GPR15 via flow cytometry resulting in mean fluorescence intensity. Data collection was planned for receptor diversity in allergen specific T cell CDR3b as compared to non-specific T cells, and TGF beta, but these data were not collected. The median value (with full range) of mean fluorescence intensity across participants is reported for each time point.
Time Frame: baseline, week 52, and week 58
Population: participants who had baseline, week 52, or week 58 Flow cytometry data
Measure: Median (Full Range); unit: mean fluorescence intensity
Arm/Group | Cashew Oral Immunotherapy | Shrimp Oral Immunotherapy | All Participants
Number analyzed (Participants) | 24 | 8 | 32
mean fluorescence intensity
  GPR15 at baseline | 1801 [0 to 39861] | 1585 [1402 to 5029] | 1664 [0 to 39861]
  GPR15 at week 52 | 1778 [0 to 10041] | 1922 [1230 to 5616] | 1798 [0 to 10041]
  GPR15 at week 58 | 1441 [0 to 33037] | 2715 [1251 to 32643] | 1609 [0 to 33037]
Statistical Analysis 1: Comparison: Cashew Oral Immunotherapy; within-group analysis of change in GPR15 from baseline to week 52; Test type: Other; p = 0.23, Mixed Models Analysis; Mean Difference (Net) = 2269
Statistical Analysis 2: Comparison: Cashew Oral Immunotherapy; within-group analysis of change in GPR15 from baseline to week 58; Test type: Other; p = 0.12, Mixed Models Analysis; Mean Difference (Net) = 1311
Statistical Analysis 3: Comparison: Cashew Oral Immunotherapy; within-group analysis of change in GPR15 from week 52 to week 58; Test type: Other; p = 0.79, Mixed Models Analysis; Mean Difference (Net) = 958
Statistical Analysis 4: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change in GPR15 from baseline to week 52; Test type: Other; p = 0.29, Mixed Models Analysis; Mean Difference (Net) = 347
Statistical Analysis 5: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change in GPR15 from baseline to week 58; Test type: Other; p = 0.29, Mixed Models Analysis; Mean Difference (Net) = 4364
Statistical Analysis 6: Comparison: Shrimp Oral Immunotherapy; within-group analysis of change in GPR15 from week 52 to week 58; Test type: Other; p = 0.42, Mixed Models Analysis; Mean Difference (Net) = 4017

ADVERSE EVENTS:
Time Frame: 64 weeks (58 weeks of OIT and food challenge plus 6 weeks follow up)
Arm/Group | Cashew Oral Immunotherapy | Shrimp Oral Immunotherapy
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/12
Other Adverse Events (participants affected / at risk) | 40/40 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cashew Oral Immunotherapy (N=40) | Shrimp Oral Immunotherapy (N=12)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cashew Oral Immunotherapy (N=40) | Shrimp Oral Immunotherapy (N=12)
Abdominal Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
ankle injury (Injury, poisoning and procedural complications) | 0 | 1
Ankles and left knee hurt when running (Injury, poisoning and procedural complications) | 1 | 0
Atopic Dermatitis Flare (Skin and subcutaneous tissue disorders) | 2 | 0
Belching (Gastrointestinal disorders) | 0 | 1
Body Soreness (General disorders) | 2 | 0
Bump on cheek (Skin and subcutaneous tissue disorders) | 1 | 0
Bump on lip (Skin and subcutaneous tissue disorders) | 1 | 0
Cervical lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Discomfort (General disorders) | 2 | 0
Ear pressure (Ear and labyrinth disorders) | 2 | 0
enlarged lymph node - status post-vaccination (Blood and lymphatic system disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 2 | 0
Photophobia (Eye disorders) | 0 | 1
Food poisoning (Injury, poisoning and procedural complications) | 1 | 0
Edema face (General disorders) | 7 | 2
Fatigue (General disorders) | 2 | 0
Fever (General disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 25 | 3
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 10 | 1
Gastroenteritis (Stomach flu) (Gastrointestinal disorders) | 1 | 1
Itchy mouth/throat/lips/tongue (Gastrointestinal disorders) | 32 | 8
Stomach pain (Gastrointestinal disorders) | 7 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 7 | 1
Heartburn (Acid Reflux) (Gastrointestinal disorders) | 1 | 0
Gum Soreness (General disorders) | 1 | 0
Hand Swelling (Vascular disorders) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 9 | 4
Wound infection (Infections and infestations) | 0 | 1
Burn (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
itchy skin (Skin and subcutaneous tissue disorders) | 2 | 0
itchy ears (Ear and labyrinth disorders) | 0 | 1
itchy eyes (Eye disorders) | 1 | 0
Itchy/Red/Eyes (Eye disorders) | 2 | 0
Jaw Tightness/Ache (Musculoskeletal and connective tissue disorders) | 0 | 1
Lightheadedness (General disorders) | 2 | 0
lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Mild conjunctival infection (Infections and infestations) | 1 | 0
Muscle Soreness (General disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 3
Agitation (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Seasonal Allergies (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema Flare (Skin and subcutaneous tissue disorders) | 5 | 2
Poison Oak (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 2
Skin Abrasion (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 7 | 4
Sour taste/reflux (Gastrointestinal disorders) | 1 | 0
Stomach Cramps due to Period (Gastrointestinal disorders) | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 3 | 0
Stomach Discomfort (No Pain) (Gastrointestinal disorders) | 7 | 1
stuffy and runny nose (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tenesmus (Gastrointestinal disorders) | 2 | 0
Throat Discomfort (Gastrointestinal disorders) | 5 | 0
Throat Discomfort, Change in Breathing (Gastrointestinal disorders) | 2 | 0
Throat Tingling (Gastrointestinal disorders) | 1 | 0
tingling sensation of mouth (Gastrointestinal disorders) | 0 | 1
TMJ (Musculoskeletal and connective tissue disorders) | 1 | 0
Tongue Tingling (Gastrointestinal disorders) | 2 | 0
Transient lesion on tongue (Gastrointestinal disorders) | 2 | 0
Transient Throat Discomfort (Gastrointestinal disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, this study did not enroll the planned number of participants and did not meet the protocol-specified threshold for statistical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT03504774/Prot_SAP_001.pdf
  • Informed Consent Form (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT03504774/ICF_000.pdf